CLINICAL TRIAL: NCT01786538
Title: Randomized Phase III Study of Oxaliplatin, Fluorouracil and Leucovorin (FOLFOX) With or Without Regorafenib in Patients With Metastatic Colorectal Cancer Progressed After First-line Irinotecan Plus Fluoropyrimidines
Brief Title: Second-line FOLFOX With or Without Regorafenib in mCRC Patients Failed to First-line Irinotecan Plus Fluoropyrimidines
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Tae Won Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Regorafenib/FOLFOX
Record Dates: First submitted 2013-02-04; First posted 2013-02-08 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; Folfox protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regorafenib/FOLFOX (Experimental)
  Interventions: Drug: Regorafenib/FOLFOX
- Placebo/FOLFOX (Active Comparator)
  Interventions: Drug: Placebo/FOLFOX

INTERVENTIONS:
Drug: Regorafenib/FOLFOX — FOLFOX consisted of oxaliplatin 85 mg/m2 on D1, leucovorin 400 mg/m2 on D1, 5-fluorouracil 400 mg/m2 intravenous bolus on D1 and 5-fluorouracil 1200 mg/m2/day continuous infusion on D1-2 (2400 mg/m2 for 46 hours). Regorafenib will be administered 160 mg/day given orally on D4-10 (7 days per each cycle of FOLFOX). Treatment will be repeated every 2 weeks and continued until disease progression, unacceptable toxicity or the patient's refusal.
  Arms: Regorafenib/FOLFOX
Drug: Placebo/FOLFOX — FOLFOX consisted of oxaliplatin 85 mg/m2 on D1, leucovorin 400 mg/m2 on D1, 5-fluorouracil 400 mg/m2 intravenous bolus on D1 and 5-fluorouracil 1200 mg/m2/day continuous infusion on D1-2 (2400 mg/m2 for 46 hours). Placebo will be administered 160 mg/day given orally on D4-10 (7 days per each cycle of FOLFOX). Treatment will be repeated every 2 weeks and continued until disease progression, unacceptable toxicity or the patient's refusal.
  Arms: Placebo/FOLFOX

SUMMARY:
Regorafenib has been proved to improved survival in patients with metastatic colorectal cancer who have been failed to all of known standard chemotherapy (The CORRECT study). The phase Ib study of regorafenib plus FOLFOX or FOLFIRI was performed and the dose of regorafenib was fixed; 160 mg/day on days 4 to 10 (7 days per cycle when combined with FOLFOX or FOLFIRI). Regorafenib plus FOLFOX as second-line chemotherapy in mCRC patients who progressed after first-line irinotecan-based chemotherapy has not been studied yet, and because there have been unmet needs for the discovery of valid targeted agent combination for the second-line FOLFOX as above reasons, the investigators planned this study of regorafenib plus FOLFOX as second-line chemotherapy in mCRC patients who progressed after first-line irinotecan-based chemotherapy.

DETAILED DESCRIPTION:
Limited active drugs are available for the treatment of patients with metastatic colorectal cancer (mCRC) at present and upfront doublet combination of fluoropyrimidines plus either oxaliplatin or irinotecan is regarded as reference strategy for patients appropriate for intensive therapy. Before the era of targeted agents, the treatment strategies in terms of either combination or sequence of cytotoxic agents were rather simple; survival outcomes did not differ according to either the administration sequence of oxaliplatin or irinotecan, or the sequential versus combination chemotherapy in the treatment continuum. However, the treatment strategies have become more complicated in the era of targeted agents.

In case of failure to first-line oxaliplatin plus fluoropyrimidines (FOLFOX or CapeOX) with or without bevacizumab, second-line chemotherapy with FOLFIRI would be administered for treatment continuum, and more various targeted agents can be combined in these setting; bevacizumab beyond progression only in patients who have been treated with first-line bevacizumab plus FOLFOX or CapeOX (TML and BRiTE), cetuximab (only for patients with wild-type KRAS), panitumumab (only for patients with wild-type KRAS), and aflibercept (VELOUR). However, there have been a few valid targeted agents which could be combined in the second line FOLFOX or CapeOX in those progressed after first-line FOLFIRI with or without targeted agents; bevacizumab beyond progression could be a valid treatment strategy only in those received first-line bevacizumab plus FOLFIRI. Higher dose of bevacizumab (10 mg/kg/2-week) could be combined to FOLFOX as second-line chemotherapy; however, it is not recommended at present in terms of cost effectiveness and higher adverse events, and cetuximab plus oxaliplatin-based chemotherapy is neither recommended by current consensus. Thus, there have been unmet needs for the discovery of valid targeted agent combination for the second-line FOLFOX as above reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the colon or the rectum.
2. Progressed during or within 6 months of first-line irinotecan plus fluoropyrimidines with or without targeted agents (bevacizumab or cetuximab).
3. Measurable or evaluable lesion(s) by RECIST 1.1.
4. Unresectable metastatic disease.
5. Age over 20 years old.
6. ECOG performance status of 1 or lower.
7. Adequate organ functions. A. Bone marrow function: ANC ≥ 1,500/mm3, platelet ≥ 100,000/mm3 B. Hepatic functions: bilirubin ≤ 1.5 X ULN, AST/ALT ≤ 2.5 X ULN (≤ 5 X ULN in cases of liver metastasis) C. Renal functions: serum Cr ≤ 1.5 X ULN or calculated CCr (Cockroft) ≥ 60 ml/min
8. Be willing and able to comply with the protocol for the duration of the study.
9. Give written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw the study at any time, without prejudice.
10. Women of childbearing potential and men must agree to use adequate contraception since signing of the IC form until at least 8 weeks after the last study drug administration.

Exclusion Criteria:

1. Prior treatment of regorafenib.
2. Prior exposure to oxaliplatin as metastatic setting is not allowed in any case; however, prior exposure to oxaliplatin as (neo)adjuvant chemo(radio)therapy is allowed if progressed after 12 months from the date of completion of oxaliplatin-containing (neo)adjuvant treatment.
3. Concurrent or previous history of another primary cancer within 3 years prior to randomisation except for curatively treated cervical cancer in situ, non-melanomatous skin cancer, superficial bladder cancer (pTis and pT1) and curatively treated thyroid cancer of any stage. Concurrent, histologically confirmed, unresected thyroid cancer without distant metastasis could be allowed with the agreement of the chief principal investigator.
4. Uncontrolled CNS metastases.
5. Prior radiation therapy would be permitted, but non-radiated evaluable lesions should be present at study entry.
6. Radiation therapy during chemotherapy is not permitted, but if the local investigator decides that radiation therapy should be given during study treatments, he should be convinced that there is no evidence of disease progression with agreement of the chief principal investigator. Radiation therapy during the chemotherapy-free interval between 1st and 2nd line chemotherapy is permitted.
7. Uncontrolled hypertension (>150/100 mmHg) despite of optimal management; anti-hypertensive drugs for BP lowering before study entry would be permitted.
8. Congestive heart failure ≥ New York Heart Association (NYHA) class 2.
9. Unstable angina, new-onset angina within 3 months, or history of myocardial infarction within 6 months before the study entry.
10. Arterial or venous thromboembolism within 6 months.
11. Serious concurrent infections or non-malignant illness.
12. Liver cirrhosis ≥ Child-Pugh class B.
13. Prior unanticipated severe toxicity to fluoropyrimidines, or known dihydropyrimidine dehydrogenase (DPD) deficiency.
14. Prior hypersensitivity to oxaliplatin (grade ≥ 2).
15. Peripheral neuropathy of grade ≥ 2.
16. Major surgery or significant traumatic injury within 28 days prior to study treatment.
17. Non-healing wound, ulcer, or bone fracture.
18. Current evidence of significant gastrointestinal bleeding or (impending) obstruction.
19. Proteinuria ≥ 3+ in the routine urinalysis; in this case, the total protein in the 24-hour urine collection should be measured, and the accrual is permitted if total protein < 3.5 g/day.
20. Concomitant participation in another clinical trial.
21. Pregnant of breast-feeding subjects. Women of child-bearing potential must have pregnancy test within 7 days and a negative result must be documented before start of study treatment.
22. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | time from randomization to disease-progression or any event (up to 1 year from the end of study treatment)

SECONDARY OUTCOMES:
Overall survival | Time from randomization to death (up to 1 year from the end of study treatment)
Response rate | every 6 weeks, up to disease progression from study treatment
Disease-control rate | every 6 weeks, up to disease progression from study treatment
  partial response + stable disease
Number of participants with adverse events | Every cycle (every 2 weeks) till the end of study treatment (because of disease progression or any event, up to 1 year)
  Adverse events will be monitored according to the NCI-CTCAE version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea